CLINICAL TRIAL: NCT05739396
Title: Effect of Core Stabalization Versus Rebound Therapy on Balance in Children With Cerebral Palsy
Brief Title: Core Stabalization and Rebound Therapy and CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, lecturer in pediatric department, faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003117
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Whole Body Vibration; Rebound Therapy; Balance; cp

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stabalization (Experimental): The core stability exercises will be used for core stabilization training of group (A) in addition to traditional physical therapy. The core stability program included 3 levels. Each exercise lasted 5 min, and the children shifted from one exercise to the next after the complete performance of the preceding exercise. The first (simple) level included supine abdominal draw-in (20 repetitions), abdominal draw-in with both knees to the chest (10-20 repetitions), and supine twist (10-20 repetitions). The second (medium) level included pelvic bridging (3e5 repetitions) and twist with a medicine ball (10e20 repetitions). Finally, the third (difficult) level included bridging with the head on a physio ball (the position was held for 3-5 s, followed by a slow relaxation phase, with 10-20 repetitions)
  Interventions: Other: core stabilization
- rebound therapy (Experimental): Rebound exercises will be applied for group B. this group will receive rebound exercise training in addition to traditional physical therapy . Rebound exercises were conducted on a mini-trampoline and BOSU ball. Passive bouncing will be conducted while the child was standing with his/her feet a shoulder-width apart. The therapist will held the child's legs while applying upward and downward movement. The bouncing started slowly. The child then will progress to include the rebound exercises, starting with active bounce, where in a hands free manner the therapist will ask the child to speed up or slow down the bounce rate according to the child's abilities
  Interventions: Other: core stabilization

INTERVENTIONS:
Other: core stabilization — The treatment session lasted one hour with short breaks of around 10 minutes and will be conducted three times per week for twelve successive weeks
  Other Names: rebound therapy

SUMMARY:
the study aims to compare the effect of core stabalization and rebound therapy on balance in children with hemiplegic cerebral palsy

DETAILED DESCRIPTION:
PURPOSE:

To compare the effect of core stabilization and rebound therapy on balance in children with hemiplegic cerebral palsy

BACKGROUND:

Cerebral palsy is primarily a disorder of movement and posture

HYPOTHESES:

There is no significant difference between core stabilization and rebound therapy on balance in children with hemiplegic cerebral palsy.

RESEARCH QUESTION:

Is there a significant difference between core stabilization and rebound therapy on balance in children with hemiplegic cerebral palsy?

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with spastic hemiplegic CP.
* Their chronological age ranged from 5 to 8 years,
* able to follow verbal commands or instructions during testing procedures,
* degree of spasticity in affected lower limbs ranged between1 to 1+ according to Modified Ashworth scale (MAS),
* they are able to understand and follow instructions given to them,

Exclusion Criteria:

* Children who had significant visual or auditory problems that may interfere with testing, - ---- patients who had contractures or fixed deformities related to the joints of the lower limbs, ---- injection with Botulinium toxin or any orthopaedic surgery in lower limbs 6m before study,
* children who were suffering from cardiopulmonary problems or epilepsy.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
balance | 12 week
  it measures the degree of tilting for each axis during dynamic conditions and calculates a medial lateral stability index (MLSI); an anterior-posteriorstability index (APSI); and an overall stability index(OSI),

SECONDARY OUTCOMES:
gross motor function measure-88 | 12 week
  measure gross motor function. higher scores indicate better outcome. scores are reported in percentage.
lafayette hand held dynamometer | 12 week
  measure isometric muscle strength of knee flexors and extensors. higher scores reflect better outcome
6 minute walk test | 12 week
  measure endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Faculty OP Therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty Of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Nemr A, Kora AN. Effect of core stabilization versus rebound therapy on balance in children with cerebral palsy. Acta Neurol Belg. 2024 Jun;124(3):843-851. doi: 10.1007/s13760-023-02430-8. Epub 2024 Jan 5. PMID 38177509